CLINICAL TRIAL: NCT05748210
Title: Development and Evaluation of a Symptom Management Mobile Health Application With Personalised Support for Children at the Early Stage of Cancer Survivorship and Their Caregivers
Brief Title: A Symptom Management Application for Children at the Early Stage of Cancer Survivorship and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Tan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PAED-2022-010
Record Dates: First submitted 2023-01-11; First posted 2023-02-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Oncology; Survivorship
Keywords: symptom management; cancer; children; caregiver; mobile health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Child-caregiver dyads in the intervention group will use the mHealth app for 12 weeks with personalised nurse support via interactive communication technologies. The design of the app will be guided by the theory of unpleasant symptoms.
  Interventions: Other: Symptom management mobile health application with personalised support
- Wait-list control group (Active Comparator): To ensure the equity of access to a potentially desirable and effective intervention (i.e., mHeath app for symptom management), participants in the wait-list control group will be invited to receive the same intervention as participants in the intervention group after the completion of all assessments on a voluntary basis.
  Interventions: Other: Wait-list Symptom management mobile health application with personalised support

INTERVENTIONS:
Other: Symptom management mobile health application with personalised support — Child-caregiver dyads in the intervention group will use the mHealth app for 12 weeks with personalised nurse support via interactive communication technologies. The design of the app will be guided by the theory of unpleasant symptoms.
  The app will comprise several interactive elements to provide children and their caregivers with real-time symptom management support. Comprehensive educational materials regarding cancer and its treatment side effects, including possible symptoms, functional limitations, and psychological responses, will be provided in the app for the children and their caregivers to gain a thorough understanding of the potential symptom burden that they may experience.
  Arms: Intervention group
Other: Wait-list Symptom management mobile health application with personalised support — To ensure the equity of access to a potentially desirable and effective intervention (i.e., mHeath app for symptom management), participants in the wait-list control group will be invited to receive the same intervention as participants in the intervention group after the completion of all assessments on a voluntary basis.
  Arms: Wait-list control group

SUMMARY:
The goal of this randomized controlled trial is to examine the efficacy of the mHealth app in improving symptoms experienced by children in the early stage of cancer survivorship, including physical function, anxiety, depressive symptoms, fatigue, peer relationships, and pain interference, and at improving the quality of life (QoL) of the children's primary caregivers

The main question it aims to answer is whether survivors who receive the symptom management mHealth app intervention will report improved symptoms, i.e., improved physical function; lower levels of anxiety, depressive symptoms, and fatigue; better peer relationships; and lower pain interference 3 months after starting the intervention. Additionally, we hypothesized that the primary caregivers (either the mother or father) would report an improved QoL 3 months after starting the intervention.

Participants in the intervention group will use the mHealth app for 12 weeks with personalised nurse support via interactive communication technologies. They are required to complete questionnaires at baseline (during medical follow-up), 1, 2, and 3 months (via electronic-based systems in the mobile app) Besides, semi-structured interviews and will be conducted to examine the usability, feasibility, and acceptability of the intervention.

DETAILED DESCRIPTION:
In Hong Kong, the incidence of paediatric cancer has been increasing in the past few years, from 180 new cancer cases in 2017 to 196 cases in 2019 [1]. The average 5-year survival rate for paediatric cancer patients is approximately 85% due to recent advances in cancer treatments [2]. The success of these treatments has resulted in a rapid growth in the population of paediatric cancer survivors globally. This population now has an average lifespan of 72 years [2]. Despite the improved survival rate, the high toxicity and low specificity of cancer treatment given at an early age induce a myriad of deleterious late effects that have a detrimental impact on survivors' physical and psychosocial well-being [3-5]. Therefore, children who have completed cancer treatment require ongoing monitoring for cancer progression and survivorship care as early as possible to manage the symptoms induced by the invasive treatment. Symptom management in paediatric oncology nursing is becoming increasingly important due to the complex treatment modalities. The benefits of effective symptom management, particularly improvements in physical functioning and reduced psychological distress, are exponential for children being treated for cancer and their caregivers throughout the cancer trajectory.

Paediatric oncology patients receive close monitoring of their somatic symptoms during their hospital stay, but there is a paucity of symptom management for children who have completed treatment and are at the early stage of survivorship. During the transition from hospital stay to home care, children and their caregivers may experience significant psychological distress due to their concerns about the child's health and uncertainties about coping with the potential symptom burden or cancer recurrence. During the first year after completing cancer treatment, many side effects related to the cancer or its treatment may persist, and other late effects may also develop [3]. The unmet needs for symptom monitoring and management for paediatric cancer survivors, particularly those in the early stage of survivorship, warrant immediate attention from healthcare professionals. It is imperative for healthcare professionals to engage in the rigorous planning, development, and implementation of appropriate interventions to support symptom management for children in the early stage of cancer survivorship and their caregivers. These interventions should be implemented at discharge to manage patient-reported symptoms and improve the children's QoL and survival rate.

Given the high utilisation of mobile technologies, integrating mobile technologies into current cancer survivorship care may be a promising and flexible approach for symptom management for children in the early stage of cancer survivorship and their caregivers. Digital health interventions have been shown to be effective at improving patient-reported outcomes in various patient populations, but there is a lack of such an intervention for paediatric cancer survivors and their caregivers to ameliorate their symptom burden in their local contexts (e.g., at home). The proposed study aims to develop a symptom management mHealth app to support children in the early stage of cancer survivorship and their caregivers and to evaluate its usability, feasibility, acceptability, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

Chinese paediatric cancer survivors will be included if they

* are aged 9 to 16 years,
* are able to read Chinese and communicate in Chinese,
* have completed active cancer treatment (within the previous 2 years), as early symptom management support is crucial to reduce the symptom burden in survivors and their caregivers throughout their survivorship, and
* have a smartphone or tablet and are willing to install the mHealth app.

The primary caregiver of the paediatric cancer survivors (either the mother or father)

* are able to read Chinese and communicate in Chinese, and
* have a smartphone or tablet and are willing to install the mHealth app with their children surviving cancer.

Exclusion Criteria:

Chinese paediatric cancer survivors will be excluded if they

* have cognitive impairments or psychiatric illnesses
* are currently participating in other symptom management studies, or
* have evidence of secondary malignancy or recurrence

The primary caregivers of the paediatric cancer survivors (either the mother or father) will be excluded if they have cognitive impairments or psychiatric illnesses.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Severity of child's symptoms | 3 months after starting the intervention
  The Chinese version of the Patient-Reported Outcomes Measurement Information System® (PROMIS-25) Pediatric-25 Profile version 2.0 is a comprehensive measure document child reports of their symptoms and functioning over the previous seven days. It comprises 24 questions and a single item on pain intensity to evaluate six domains, including physical function, anxiety, depressive symptoms, fatigue, peer relationship, and pain interference. Each domain has Each item has a 5-point Likert scale ranging from ''never'' to ''almost always'' in most domains and from ''with no trouble'' to ''not able to do'' for the physical functioning domain. Higher scores indicate more of the measured symptom being experienced, which signifies worse functioning for anxiety, depression, fatigue, and pain interference, and better physical functioning, and peer relationships.

SECONDARY OUTCOMES:
Severity of child's symptoms | 1 and 2 months after starting the intervention
  The Chinese version of the Patient-Reported Outcomes Measurement Information System® (PROMIS-25) Pediatric-25 Profile version 2.0 is a comprehensive measure document child reports of their symptoms and functioning over the previous seven days. It comprises 24 questions and a single item on pain intensity to evaluate six domains, including physical function, anxiety, depressive symptoms, fatigue, peer relationship, and pain interference. Each domain has Each item has a 5-point Likert scale ranging from ''never'' to ''almost always'' in most domains and from ''with no trouble'' to ''not able to do'' for the physical functioning domain. Higher scores indicate more of the measured symptom being experienced, which signifies worse functioning for anxiety, depression, fatigue, and pain interference, and better physical functioning, and peer relationships.
Caregivers' quality of life | 1, 2 and 3 months after starting the intervention
  Primary caregivers' quality of life will be assessed using the Chinese version of the World Health Organization's Quality of Life Instrument at baseline and 3 months after starting the intervention. It is a generic health status measure in assessing the overall QoL and general health (2 items), physical health (7 items), psychological health (6 items), social relationships (3 items), and environment (8 items) using a five-point Likert scale. The item scores were added to calculate the domain scores, where a higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ankie Tan Cheung, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No